CLINICAL TRIAL: NCT01014494
Title: A Randomized, Double Blind Clinical Investigation to Evaluate the Safety, Tolerability, and Preliminary Performance of Adaprev™ in Improving Recovery of Tendon Function in Subjects Undergoing Surgical Repair of Flexor Tendons in Zone II of the Hand
Brief Title: Adaprev in Digital Flexor Tendon Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renovo (Industry)
Responsible Party: Harriet Wibberley, Senior Clinical Project Manager, Renovo
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: RN1008-0083
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Tendon Injuries
MeSH Terms: conditions — Tendon Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active - Adaprev (Experimental): Adaprev (Class III medical device)
  Interventions: Device: Adaprev
- Standard Care (No Intervention): No different treatment to normal

INTERVENTIONS:
Device: Adaprev — Class III Medical Device
  Other Names: Product contains mannose-6-phosphate
  Arms: Active - Adaprev

SUMMARY:
This study is being undertaken to verify the safety and performance of Adaprev™, a Class III medical device, when administered as a short term implant into the tendon sheath at the time of surgery, on the post-operative function of severed digital tendons. Subjects are randomised to either Adaprev or standard care and attend visits for 26 weeks following surgery. This clinical investigation will recruit 44 subjects in the UK at up to 10 clinical trial sites.

ELIGIBILITY:
Inclusion Criteria:

- Subjects aged 18 years and above with complete division of the Flexor Digitorum Profundus (FDP) tendon in Zone II.

Exclusion Criteria:

* Subjects with additional complicated injuries
* Subjects whose flexor tendon repair involves a finger with less than full tendon function prior to the injury requiring repair
* Subjects who are undergoing surgical repair of the severed tendon(s) more than four days after the injury occurred.
* Subjects with a history of clinical significant hypersensitivity to any of the devices, drugs or surgical dressings to be used in this trial.
* Subjects with conditions which may delay healing.
* Subjects who are taking, or have taken, any investigational drugs within 3 months prior to the screening visit.
* Females who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The primary trial endpoint will be the assessment of safety and local tolerability for a period up to twenty six weeks after dosing. | 26 weeks post surgery

SECONDARY OUTCOMES:
The secondary endpoint will be an evaluation of the performance of Adaprev™ as measured by the range of motion of the treated finger at twenty six weeks after tendon repair | 26 weeks post surgery

CONTACTS AND LOCATIONS:
Overall Officials: John Hutchison, MBBS PhD, Study Director — Renovo Ltd
Locations (9):
- United Kingdom (9):
  - Mr P Gillespie, Addenbrooke's Hospital, Cambridge, Cambridge
  - University Hospital of South Manchester NHS Foundation Trust, Manchester, Greater Manchester
  - Mr F Schreuder, The Lister Hospital, Stevenage, Hertfordshire
  - Royal London Hospital, Barts and The London Hospital, London, London
  - Royal Free Hospital, London, London
  - Chelsea & Westminster Hospital, London, London
  - Mr R Dunn, Salisbury District Hospital, Salisbury
  - Mr D Warwick, Southampton General Hospital, Southampton
  - Abertawe Bro Morgannwg University Nhs Trust, Swansea